CLINICAL TRIAL: NCT05472077
Title: Saliva Testing for SARS-CoV-2 With Lollipop Swab
Brief Title: Lollipop COVID-19 Testing Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues with the Enrollment Location
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-1011; A536756 (Other: UW Madison); SMPH\PEDIATRICS\INFECT DIS (Other: UW Madison); Protocol Version 07/15/2022 (Other: UW Madison)
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; SARS CoV 2 Infection; COVID-19 Pandemic
Keywords: saliva collection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with COVID-19 Symptom(s) (Experimental): Participants 4 years old or older with at least one COVID-19 symptom being tested for the virus
  Interventions: Diagnostic Test: Lollipop Swab

INTERVENTIONS:
Diagnostic Test: Lollipop Swab — The "lollipop" swab is a typical swab that would be used to obtain routine pharyngeal samples. Participants are instructed to suck on the swab for 20 second, as they would suck on a lollipop.

SUMMARY:
This study will explore whether lollipop swabs are more acceptable and perform as well as nasal swabs with PCR testing. The study will be open to enrollment for both children and adults in the Madison community who have at least one COVID-19 symptom that has presented in the last 5 days and who have not had a positive COVID-19 test for a previous illness within the past 3 months. Participants can expect to be in the study for the duration of the swabbing, approximately 10 minutes.

DETAILED DESCRIPTION:
This study will test the hypothesis that lollipop swabs are more acceptable to individuals and PCR testing is non-inferior to performing PCR on nasal swabs. To test this hypothesis, the study team will work with local community testing sites to incorporate a lollipop swab for PCR at the time a symptomatic individual receives a nasal swab for PCR that is part of the DHS program. The study will address the following two key questions:

1. Are lollipop swabs more acceptable to individuals when compared to nasal swabs?
2. Will lollipop swabs perform as well as nasal swabs with PCR-based testing?

Participants with at least one COVID-19 symptom will be asked to suck on a swab for 20 seconds, like sucking on a lollipop. They then will be asked which COVID-19 PCR testing they would prefer if they had to do the testing again, nasal PCR versus lollipop PCR.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 years or above
* Have at least one COVID-19 symptom that has presented in the last 5 days and will undergo a nasal PCR test at a local community testing site

Exclusion Criteria:

* Positive COVID-19 test in the past 3 months for a previous illness

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Participant Sample Collection Preference | Day 1 (up to 10 minutes)
  The acceptance of the lollipop swab relative to nasal swab collection will be measured by asking participants which sample collection method they prefer. Count of participants for each sample collection method will be reported.
Number of Positive COVID-19 Diagnoses | Day 1 (up to 10 minutes)
  The investigators will compare results of the lollipop swab and nasal swab to assess the efficacy of the lollipop swab to diagnose COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Wald, MD, Principal Investigator — University of Wisconsin, Madison; Shelby O'Connor, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No